CLINICAL TRIAL: NCT06192498
Title: Comparison of the Effectiveness of Virtual Reality Glasses, Kaleidoscope and Distraction Cards in Reducing Pain and Anxiety During Blood Draw in Children: A Randomized Controlled Study
Brief Title: Effects of Virtual Reality Glasses, Kaleidoscope and Distraction Cards on Pain and Anxiety During Blood Draw in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-2018/22
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Acute Pain; Virtual Reality; Kaleidoscope; Distraction Cards; Nursing Caries; Children, Only; Fear; Anxiety
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality Glasses Group (Experimental): Virtual Reality(VR) Glasses were introduced to the children pre-procedure. The children were made to watch a video with VR glasses before starting the application and it continued until the end of the Blood Draw procedure.
  Interventions: Other: Virtual Reality Glasses
- Kaleidoscope Group (Experimental): Kaleidoscope were introduced to the children pre-procedure. The children were made to watch Kaleidoscope before starting the application and it continued until the end of the Blood Draw procedure.
  Interventions: Other: Kaleidoscope
- Distraction Cards Group (Experimental): Distraction Cards were introduced to the children pre-procedure. The children were made to apply Distraction Cards before starting the application and it continued until the end of the Blood Draw procedure.
  Interventions: Other: Distraction Cards
- Control Group (No Intervention): In this group, children received routine blood draw procedure.

INTERVENTIONS:
Other: Virtual Reality Glasses — Virtual Reality(VR) Glasses were introduced to the children pre-procedure. The children were made to watch a video with VR glasses before starting the application and it continued until the end of the Blood Draw procedure.
  Arms: Virtual Reality Glasses Group
Other: Kaleidoscope — Kaleidoscope were introduced to the children pre-procedure. The children were made to watch Kaleidoscope before starting the application and it continued until the end of the Blood Draw procedure.
  Arms: Kaleidoscope Group
Other: Distraction Cards — Distraction Cards were introduced to the children pre-procedure. The children were made to apply Distraction Cards before starting the application and it continued until the end of the Blood Draw procedure.
  Arms: Distraction Cards Group

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of distraction by using Virtual Reality Glasses, Kaleidoscope and Distraction Cards in reducing pain and anxiety during blood draw in children.

DETAILED DESCRIPTION:
n the literature, it is stated that nurses should use pharmacological and non-pharmacological methods in pain and anxiety management in painful procedures. Evidence-based studies are needed to show the effectiveness of non-pharmacological methods in reducing pain during invasive procedures and to investigate the effects of easy-to-apply methods on pain. In light of this information, this study aimed to compare the effect of distraction by using Virtual Reality Glasses, Kaleidoscope and Distraction Cards in reducing pain and anxiety during blood draw in children.

This study is a prospective, randomized and controlled trial. Children aged 7 to 11 years who required blood draw were divided into three groups; Virtual Reality Glasses, Kaleidoscope, Distraction Cards and Control. Data were obtained through face-to-face interviews with the children, their parents, and the observer before and after the procedure. The children's pain levels were assessed and reported by the parents and observers and the children themselves who self-reported using Wong-Baker FACES. The children's anxiety levels were also assessed using the Children's Fear Scale.

The study population consisted of children aged 7 to 11 years who presented to the children's blood draw room of the hospital.

Sample of the study consisted of a total of 400 children who met the sample selection criteria and were selected via randomization method.

Children were randomized into three groups: Virtual Reality Glasses group (n= 100), Kaleidoscope group (n= 100), Distraction Cards group (n= 100) and Control group (n= 100).

Data were collected using the Interview and Observation Form, Wong-Baker FACES Pain Rating Scale, Children's Fear Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7-11,
* Volunteering of the child and parent to participate in the study,
* Blood draw for routine control purposes,
* Blood draw should be done by the same nurse,
* The needle on which blood draw will be performed must be of the same thickness.

Exclusion Criteria:

* The child has any acute or chronic disease,
* The child has a mental disability, vision, speech or communication problems,
* The parent has hearing, vision or verbal communication difficulties,
* The child used analgesics in the last 6 hours,
* Infection, disruption of skin integrity and rash in the area where the application will be made,
* Exclusion criteria were that the parent or child wanted to leave the study at any point.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Wong-Baker FACES Pain Rating Scale | Through painful procedure completion, an average of 10 minutes
  In the study, pain level evaluations, the children's self-evaluations, parents' evaluations and the researcher's evaluations were carried out using the WB-FACES scale. This scale was developed by Donna Wong and Connie Morain Baker in 1988. The scale is graded between 0-10 points. A smiling face on the far left symbolizes "no pain" (0 very happy/no pain) and the pain increases from left to right. On the other hand, a crying face on the far right symbolizes "unbearable pain" (10 'hurts worst'). As the numbers increase in this scoring system, facial expressions also change referring to an increase in pain levels.
Children's Fear Scale | Through painful procedure completion, an average of 10 minutes
  CFS is used for measuring the child's anxiety level. CFS is a scale which makes an evaluation from 0 to 4 consisting of five facial expressions drawn to show expressions that vary from neutral expression (0=no anxiety) to scared face (4=severe anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, PhD., Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Karaman Education and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Ates Besirik S, Canbulat Sahiner N. Comparison of the effectiveness of three different distraction methods in reducing pain and anxiety during blood drawing in children: A randomized controlled study. J Pediatr Nurs. 2024 Nov-Dec;79:225-233. doi: 10.1016/j.pedn.2024.09.009. Epub 2024 Sep 19. PMID 39303378